CLINICAL TRIAL: NCT00246012
Title: A Phase 1/2, Multi-Center, Blinded, Randomized, Controlled Study of the Safety and Efficacy of the Human Monoclonal Antibody to Human α ν Integrins (CNTO 95), Alone and in Combination With Dacarbazine, in Subjects With Stage IV Melanoma
Brief Title: A Safety and Efficacy Study of Intetumumab, Alone and in Combination With Dacarbazine, in Participants With Stage 4 Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Collaborators: Janssen-Cilag Farmaceutica, S.R.L. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR006004; C1034T02 (Other: Centocor, Inc); 2004-002130-18 (EudraCT Number)
Record Dates: First submitted 2005-10-28; First posted 2005-10-31 (Estimated); Results first posted 2013-08-19 (Estimated); Last update posted 2013-08-19 (Estimated); Status verified 2013-07

CONDITIONS: Melanoma
Keywords: Melanoma; Neoplasm; CNTO 95; Dacarbazine; Intetumumab
MeSH Terms: conditions — Melanoma; Neoplasms | interventions — intetumumab; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Intetumumab 3 mg/kg [Phase 1 (Part 1)] (Experimental): Intetumumab will be administered at the dose of 3 milligram per kilogram (mg/kg) as intravenous infusion (a fluid or a medicine delivered into a vein by way of a needle) over a period of 2 hours (hr) (± 15 minutes) once every 3 weeks until the occurrence of dose limiting toxicities (DLTs). If after an evaluation of the preliminary single-dose pharmacokinetics, receptor saturation is not observed at the 3 mg/kg or 5 mg/kg dose level, that dose of intetumumab will be discontinued in Part 1 and participants will be treated at the highest, documented safe dose level at which receptor saturation is observed.
  Interventions: Drug: Intetumumab
- Intetumumab 5 mg/kg [Phase 1 (Part 1)] (Experimental): Intetumumab will be administered at the dose of 5 mg/kg as intravenous infusion over a period of 2 hr (± 15 minutes) once every 3 weeks until the occurrence of DLTs. If after an evaluation of the preliminary single-dose pharmacokinetics, receptor saturation is not observed at the 3 mg/kg or 5 mg/kg dose level, that dose of intetumumab will be discontinued in Part 1 and participants will be treated at the highest, documented safe dose level at which receptor saturation is observed.
  Interventions: Drug: Intetumumab
- Intetumumab 10 mg/kg [Phase 1 (Part 1)] (Experimental): Intetumumab will be administered at the dose of 10 mg/kg as intravenous infusion over a period of 2 hr (± 15 minutes) once every 3 weeks until the occurrence of DLTs.
  Interventions: Drug: Intetumumab
- Dacarbazine + intetumumab 5 mg/kg [Phase 1 (Part 2)] (Experimental): Intetumumab will be administered at the dose of 5 mg/kg as intravenous infusion over a period of 2 hr (± 15 minutes) once every 3 weeks for 8 cycles until no evidence of disease progression or unacceptable toxicity. If participants respond to therapy with stable disease (SD) or better, they will be considered eligible to receive up to 8 cycles of extended administrations. Commercially available dacarbazine will be administered at the dose of 1000 milligram per meter-square (mg/m^2) intravenously over a period of 60 minutes (± 30 minutes) prior to intetumumab infusion.
  Interventions: Drug: Intetumumab; Drug: Dacarbazine
- Dacarbazine + intetumumab 10 mg/kg [Phase 1 (Part 2)] (Experimental): Intetumumab will be administered at the dose of 10 mg/kg as intravenous infusion over a period of 2 hr (± 15 minutes) once every 3 weeks for 8 cycles until no evidence of disease progression or unacceptable toxicity. If participants respond to therapy with SD or better, they will be considered eligible to receive up to 8 cycles of extended administrations. Commercially available dacarbazine will be administered at the dose of 1000 mg/m^2 intravenously over a period of 60 minutes (± 30 minutes) prior to intetumumab infusion.
  Interventions: Drug: Intetumumab; Drug: Dacarbazine
- Dacarbazine + placebo [Phase 2] (Experimental): Placebo will be administered intravenously over a period of 2 hr (±15 minutes). Commercially available dacarbazine will be administered at the dose of 1000 mg/m^2 intravenously over a period of 60 minutes (± 30 minutes) prior to placebo infusion. In case participants are unable to tolerate dacarbazine even after 2 dose reductions, they will be given the option to continue with 10 mg/kg intetumumab alone.
  Interventions: Drug: Dacarbazine; Drug: Placebo
- Intetumumab 5 mg/kg [Phase 2] (Experimental): Intetumumab will be administered at the dose of 5 mg/kg as intravenous infusion over a period of 2 hr (± 15 minutes) once every 3 weeks for 8 cycles until no evidence of disease progression or unacceptable toxicity. If participants respond to therapy with SD or better, they are considered eligible to receive up to 8 cycles of extended administrations.
  Interventions: Drug: Intetumumab
- Intetumumab 10 mg/kg [Phase 2] (Experimental): Intetumumab will be administered at the dose of 10 mg/kg as intravenous infusion over a period of 2 hr (± 15 minutes) once every 3 weeks for 8 cycles until no evidence of disease progression or unacceptable toxicity. If participants respond to therapy with SD or better, they are considered eligible to receive up to 8 cycles of extended administrations.
  Interventions: Drug: Intetumumab
- Dacarbazine + intetumumab 10 mg/kg [Phase 2] (Experimental): Intetumumab will be administered at the dose of 10 mg/kg as intravenous infusion over a period of 2 hr (± 15 minutes) once every 3 weeks for 8 cycles until no evidence of disease progression or unacceptable toxicity. If participants respond to therapy with SD or better, they are considered eligible to receive up to 8 cycles of extended administrations. Commercially available dacarbazine will be administered at the dose of 1000 mg/m^2 intravenously over a period of 60 minutes (± 30 minutes) prior to intetumumab infusion.
  Interventions: Drug: Intetumumab; Drug: Dacarbazine

INTERVENTIONS:
Drug: Intetumumab — Intetumumab will be administered at the dose of 3 milligram per kilogram (mg/kg) as intravenous infusion (a fluid or a medicine delivered into a vein by way of a needle) over a period of 2 hours (hr) (± 15 minutes) once every 3 weeks until the occurrence of dose limiting toxicities (DLTs). In Phase 2, intetumumab (5 mg/kg or 10 mg/kg) will be administered for 8 cycles until no evidence of disease progression or unacceptable toxicity. If a participant responds to therapy with stable disease (SD) or better, the participant will be eligible to receive up to 8 cycles of extended administrations.
  Arms: Dacarbazine + intetumumab 10 mg/kg [Phase 1 (Part 2)]; Dacarbazine + intetumumab 10 mg/kg [Phase 2]; Dacarbazine + intetumumab 5 mg/kg [Phase 1 (Part 2)]; Intetumumab 10 mg/kg [Phase 1 (Part 1)]; Intetumumab 10 mg/kg [Phase 2]; Intetumumab 3 mg/kg [Phase 1 (Part 1)]; Intetumumab 5 mg/kg [Phase 1 (Part 1)]; Intetumumab 5 mg/kg [Phase 2]
Drug: Dacarbazine — Commercially available dacarbazine will be administered intravenously over a 60-minute period (+30 minutes/-30 minutes) and prior to the intetumumab/placebo infusion. In case participants are unable to tolerate dacarbazine even after 2 dose reductions, they will be given the option to continue on intetumumab alone.
  Arms: Dacarbazine + intetumumab 10 mg/kg [Phase 1 (Part 2)]; Dacarbazine + intetumumab 10 mg/kg [Phase 2]; Dacarbazine + intetumumab 5 mg/kg [Phase 1 (Part 2)]; Dacarbazine + placebo [Phase 2]
Drug: Placebo — Placebo will be administered intravenously over a period of 2 hours (+15 minutes/-15 minutes).
  Arms: Dacarbazine + placebo [Phase 2]

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the intetumumab, alone and in combination with dacarbazine, in patients with stage 4 melanoma.

DETAILED DESCRIPTION:
This is a Phase 1/2, multi-center, randomized (the study medication is assigned by chance) study. This study will be conducted in 2 Phases (Phase 1 and Phase 2). Phase 1 of this study will be non-randomized, open-label (all people know the identity of the intervention) and dose-escalation phase. It includes screening period and treatment period, which consists of 2 parts (Part 1 and Part 2). In Part 1, participants will receive 1 of 3 single dose levels of intetumumab [3 milligram per kilogram (mg/kg), 5 mg/kg or 10 mg/kg]. Part 2 will include 2 dose cohorts: dacarbazine plus intetumumab (5 mg/kg) or dacarbazine plus intetumumab (10 mg/kg). Phase 2 of this study will be randomized, blinded (neither physician nor participant knows the intervention which the participant will receive) and controlled (an inactive substance and other medication is compared with a study medication to test whether the medication has a real effect in this clinical study). This phase of the study will include screening period, treatment period (8 cycles of treatment with every cycle once in 3 weeks) and follow-up period (24 weeks). During the treatment period, participants will be randomly assigned to 1 of 4 treatment groups, Group 1: dacarbazine plus placebo, Group 2: intetumumab (5 mg/kg), Group 3: intetumumab (10 mg/kg) and Group 4: dacarbazine plus intetumumab. Randomization will be further based on the site of metastases and Eastern Cooperative Oncology Group performance status at Baseline. Single-medication intetumumab treatment groups will be open-label, while the dacarbazine plus intetumumab or placebo groups will be blinded. The total duration of the Phase 2 of this study will be up to 52 weeks or up to 76 weeks in case of extended dosing (extended administrations [up to 8 additional cycles] of the same assigned treatment will be allowed for participants that are responding to therapy with stable disease or better). Participants will be assessed for incidence of dose limiting toxicities, pharmacokinetics and tumor responses. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed melanoma including ocular and mucosal
* Documented AJCC (American Joint Committee on Cancer) Stage 3 unresectable or Stage 4 melanoma (Phase 1); AJCC Stage 4 melanoma (Phase 2)
* Radiographically measurable disease or measurable skin lesions
* Prior chemotherapy for metastatic melanoma will be allowed for Phase 1, while previously untreated for melanoma by chemotherapy will be allowed for Phase 2
* Agrees to protocol-defined use of effective contraception

Exclusion Criteria:

* History of receiving murine or human/murine recombination products of human αν integrins
* Known human immunodeficiency virus (HIV) positivity and clinically important active infection
* Presence of bone metastases or malignant effusions (non-measurable lesions) and central nervous system metastases
* Prior radiation to target lesions
* Concurrent immunotherapy, biotherapy, radiotherapy, chemotherapy, or investigational therapy and therapeutic use of anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2005-05; Primary Completion 2008-06 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.
Locations (32):
- United States (17):
  - Scottsdale, Arizona
  - La Jolla, California
  - Santa Monica, California
  - Walnut Creek, California
  - Aurora, Colorado
  - Washington D.C., District of Columbia
  - Miami, Florida
  - Atlanta, Georgia
  - Park Ridge, Illinois
  - Beech Grove, Indiana
  - Omaha, Nebraska
  - Buffalo, New York
  - New York, New York
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Dallas, Texas
  - Seattle, Washington
- Germany (10):
  - Berlin
  - Bonn
  - Buxtehude
  - Düsseldorf
  - Essen
  - Hanover
  - Jena
  - Kiel
  - Mannheim
  - Münster
- United Kingdom (5):
  - Cambridge
  - London
  - Manchester
  - Sheffield
  - Southampton

RESULTS

PARTICIPANT FLOW:
Groups:
- Intetumumab 3 mg/kg [Phase 1 (Part 1)]: Intetumumab was administered at the dose of 3 milligram per kilogram (mg/kg) as intravenous infusion (a fluid or a medicine delivered into a vein by way of a needle) over a period of 2 hours (hr) (± 15 minutes) once every 3 weeks until the occurrence of dose limiting toxicities (DLTs). If after an evaluation of the preliminary single-dose pharmacokinetics, receptor saturation was not observed at the 3 mg/kg or 5 mg/kg dose level, that dose of intetumumab was discontinued in Part 1 and participants were treated at the highest, documented safe dose level at which receptor saturation was observed.
- Intetumumab 5 mg/kg [Phase 1 (Part 1)]: Intetumumab was administered at the dose of 5 mg/kg as intravenous infusion over a period of 2 hr (± 15 minutes) once every 3 weeks until the occurrence of DLTs. If after an evaluation of the preliminary single-dose pharmacokinetics, receptor saturation was not observed at the 3 mg/kg or 5 mg/kg dose level, that dose of intetumumab was discontinued in Part 1 and participants were treated at the highest, documented safe dose level at which receptor saturation was observed.
- Intetumumab 10 mg/kg [Phase 1 (Part 1)]: Intetumumab was administered at the dose of 10 mg/kg as intravenous infusion over a period of 2 hr (± 15 minutes) once every 3 weeks until the occurrence of DLTs.
- Dacarbazine + Intetumumab 5 mg/kg [Phase 1 (Part 2)]: Intetumumab was administered at the dose of 5 mg/kg as intravenous infusion over a period of 2 hr (± 15 minutes) once every 3 weeks for 8 cycles until no evidence of disease progression or unacceptable toxicity. If participants responded to therapy with stable disease (SD) or better, they were considered eligible to receive up to 8 cycles of extended administrations. Commercially available dacarbazine was administered at the dose of 1000 milligram per meter-square (mg/m^2) intravenously over a period of 60 minutes (± 30 minutes) prior to intetumumab infusion.
- Dacarbazine + Intetumumab 10 mg/kg [Phase 1 (Part 2)]; Dacarbazine + Intetumumab 10 mg/kg [Phase 2]: Intetumumab was administered at the dose of 10 mg/kg as intravenous infusion over a period of 2 hr (± 15 minutes) once every 3 weeks for 8 cycles until no evidence of disease progression or unacceptable toxicity. If participants responded to therapy with SD or better, they were considered eligible to receive up to 8 cycles of extended administrations. Commercially available dacarbazine was administered at the dose of 1000 mg/m^2 intravenously over a period of 60 minutes (± 30 minutes) prior to intetumumab infusion.
- Dacarbazine + Placebo [Phase 2]: Placebo was administered intravenously over a period of 2 hr (±15 minutes). Commercially available dacarbazine was administered at the dose of 1000 mg/m^2 intravenously over a period of 60 minutes (± 30 minutes) prior to placebo infusion. In case participants were unable to tolerate dacarbazine even after 2 dose reductions, they were given the option to continue with 10 mg/kg intetumumab alone.
- Intetumumab 5 mg/kg [Phase 2]: Intetumumab was administered at the dose of 5 mg/kg as intravenous infusion over a period of 2 hr (± 15 minutes) once every 3 weeks for 8 cycles until no evidence of disease progression or unacceptable toxicity. If participants responded to therapy with SD or better, they were considered eligible to receive up to 8 cycles of extended administrations.
- Intetumumab 10 mg/kg [Phase 2]: Intetumumab was administered at the dose of 10 mg/kg as intravenous infusion over a period of 2 hr (± 15 minutes) once every 3 weeks for 8 cycles until no evidence of disease progression or unacceptable toxicity. If participants responded to therapy with SD or better, they were considered eligible to receive up to 8 cycles of extended administrations.
Period: Overall Study
Arm/Group | Intetumumab 3 mg/kg [Phase 1 (Part 1)] | Intetumumab 5 mg/kg [Phase 1 (Part 1)] | Intetumumab 10 mg/kg [Phase 1 (Part 1)] | Dacarbazine + Intetumumab 5 mg/kg [Phase 1 (Part 2)] | Dacarbazine + Intetumumab 10 mg/kg [Phase 1 (Part 2)] | Dacarbazine + Placebo [Phase 2] | Intetumumab 5 mg/kg [Phase 2] | Intetumumab 10 mg/kg [Phase 2] | Dacarbazine + Intetumumab 10 mg/kg [Phase 2]
Started | 3 | 3 | 3 | 3 | 3 | 32 | 32 | 33 | 32
Treated | 3 | 3 | 3 | 3 | 3 | 31 | 31 | 33 | 32
Completed | 0 | 2 | 1 | 0 | 0 | 4 | 1 | 5 | 4
Not Completed | 3 | 1 | 2 | 3 | 3 | 28 | 31 | 28 | 28
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Disease progression | 3 | 1 | 2 | 3 | 3 | 25 | 30 | 27 | 26
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Randomly assigned but not treated | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intetumumab 3 mg/kg [Phase 1 (Part 1)] | Intetumumab 5 mg/kg [Phase 1 (Part 1)] | Intetumumab 10 mg/kg [Phase 1 (Part 1)] | Dacarbazine + Intetumumab 5 mg/kg [Phase 1 (Part 2)] | Dacarbazine + Intetumumab 10 mg/kg [Phase 1 (Part 2)] | Dacarbazine + Placebo [Phase 2] | Intetumumab 5 mg/kg [Phase 2] | Intetumumab 10 mg/kg [Phase 2] | Dacarbazine + Intetumumab 10 mg/kg [Phase 2] | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 31 | 31 | 33 | 32 | 142
Age Continuous [Mean (Standard Deviation); unit: Years] | 62.0 (10.82) | 46.7 (6.66) | 61.7 (11.59) | 52.7 (15.01) | 66.0 (18.73) | 63.5 (14.17) | 67.3 (11.44) | 61.5 (12.39) | 57.2 (11.45) | 61.8 (12.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 1 | 1 | 13 | 8 | 7 | 14 | 47
  Male | 2 | 2 | 2 | 2 | 2 | 18 | 23 | 26 | 18 | 95
Region of Enrollment [Number; unit: Participants]
  Germany | 0 | 0 | 0 | 0 | 0 | 9 | 12 | 10 | 13 | 44
  United Kingdom | 0 | 0 | 0 | 0 | 0 | 6 | 9 | 4 | 5 | 24
  United States | 3 | 3 | 3 | 3 | 3 | 16 | 10 | 19 | 14 | 74

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) - Phase 1
Description: The DLT is defined as any Grade 3 or higher adverse event identified by the safety data monitoring committee as attributable to intetumumab except for hypersensitivity reactions, which are not considered DLTs unless there are 2 or more occurrences of greater than or equal to Grade 3 hypersensitivity reaction within a group.
Time Frame: Up to 21 days post-first infusion from the last treated participant in Phase 1
Population: Safety population included all the participants who received at least 1 (partial or complete) dose of intetumumab/placebo or dacarbazine.
Measure: Number; unit: Participants
Arm/Group | Intetumumab 3 mg/kg [Phase 1 (Part 1)] | Intetumumab 5 mg/kg [Phase 1 (Part 1)] | Intetumumab 10 mg/kg [Phase 1 (Part 1)] | Dacarbazine + Intetumumab 5 mg/kg [Phase 1 (Part 2)] | Dacarbazine + Intetumumab 10 mg/kg [Phase 1 (Part 2)]
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Maximum Observed Serum Concentration (Cmax) of Intetumumab - Phase 1 (Part 1)
Description: The maximum observed analyte concentration in serum was reported.
Time Frame: Pre-infusion, post-infusion at 2, 4, 8, 24 hour, Day 8, Day 15, post-last dose (3 weeks or 1 week) and 3 months post-last dose
Population: The Pharmacokinetics (PK)-evaluable population included all the participants who had at least 1 PK sample and who received at least 1 (partial or complete) dose of intetumumab.
Measure: Mean (Standard Deviation); unit: Microgram per milliliter (mcg/mL)
Arm/Group | Intetumumab 3 mg/kg [Phase 1 (Part 1)] | Intetumumab 5 mg/kg [Phase 1 (Part 1)] | Intetumumab 10 mg/kg [Phase 1 (Part 1)]
Number analyzed (Participants) | 3 | 3 | 3
Microgram per milliliter (mcg/mL) | 94.44 (9.037) | 199.45 (64.093) | 306.86 (54.979)

3. Primary Outcome: Area Under the Serum Concentration Versus Time Curve (AUC) of Intetumumab - Phase 1 (Part 1)
Description: The AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption.
Time Frame: as for outcome 2
Population: The PK-evaluable population included all the participants who had at least 1 PK sample and who received at least 1 (partial or complete) dose of intetumumab. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: mcg*day/mL
Arm/Group | Intetumumab 3 mg/kg [Phase 1 (Part 1)] | Intetumumab 5 mg/kg [Phase 1 (Part 1)] | Intetumumab 10 mg/kg [Phase 1 (Part 1)]
Number analyzed (Participants) | 1 | 1 | 3
mcg*day/mL | 257.55 (NA) — Standard deviation was not estimable based on one subject. | 503.71 (NA) — Standard deviation was not estimable based on one subject. | 1479.07 (149.851)

4. Primary Outcome: Half-life of Intetumumab - Phase 1 (Part 1)
Description: Plasma decay half-life is the time measured for the plasma concentration of the drug to decrease by one half.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Intetumumab 3 mg/kg [Phase 1 (Part 1)] | Intetumumab 5 mg/kg [Phase 1 (Part 1)] | Intetumumab 10 mg/kg [Phase 1 (Part 1)]
Number analyzed (Participants) | 1 | 1 | 3
Days | 2.03 (NA) — Standard deviation was not estimable based on one subject. | 2.13 (NA) — Standard deviation was not estimable based on one subject. | 5.33 (1.001)

5. Primary Outcome: Total Clearance (CL) of Intetumumab After Intravenous Administration - Phase 1 (Part 1)
Description: The CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/day/kg
Arm/Group | Intetumumab 3 mg/kg [Phase 1 (Part 1)] | Intetumumab 5 mg/kg [Phase 1 (Part 1)] | Intetumumab 10 mg/kg [Phase 1 (Part 1)]
Number analyzed (Participants) | 1 | 1 | 3
mL/day/kg | 11.85 (NA) — Standard deviation was not estimable based on one subject. | 9.96 (NA) — Standard deviation was not estimable based on one subject. | 6.79 (1.634)

6. Primary Outcome: Volume of Distribution (Vz) of Intetumumab - Phase 1 (Part 1)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | Intetumumab 3 mg/kg [Phase 1 (Part 1)] | Intetumumab 5 mg/kg [Phase 1 (Part 1)] | Intetumumab 10 mg/kg [Phase 1 (Part 1)]
Number analyzed (Participants) | 1 | 1 | 3
mL/kg | 34.69 (NA) — Standard deviation was not estimable based on one subject. | 30.63 (NA) — Standard deviation was not estimable based on one subject. | 50.80 (4.981)

7. Primary Outcome: Accumulation Ratio (R) of Intetumumab - Phase 1 (Part 1)
Description: The R is obtained by dividing AUC at two different time points.
Time Frame: as for outcome 2
Population: The PK-evaluable population included all the participants who had at least 1 PK sample and who received at least 1 (partial or complete) dose of intetumumab. Serum concentration data was insufficient to robustly estimate the accumulation ratio.
Arm/Group | Intetumumab 3 mg/kg [Phase 1 (Part 1)] | Intetumumab 5 mg/kg [Phase 1 (Part 1)] | Intetumumab 10 mg/kg [Phase 1 (Part 1)]
Number analyzed (Participants) | 0 | 0 | 0

8. Primary Outcome: Progression-Free Survival (PFS) - Phase 2
Description: The PFS was defined as the time from the date of randomization to the date of initial documented progressive disease (PD), or the date of initial documented symptomatic deterioration, or the date of death, whichever occurred first. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as at least a 20% increase in the sum of the longest diameter of target lesions, taking as a reference the smallest sum longest diameter recorded since the treatment started or the appearance of 1 or more new lesions.
Time Frame: From the date of randomization to date of initial documented progressive disease or death, whichever occured first, as assessed upto 6 months after last dose of study medication
Population: The Intent-to-treat (ITT) population included all the participants who were randomly assigned to treatment.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Dacarbazine + Placebo [Phase 2] | Intetumumab 5 mg/kg [Phase 2] | Intetumumab 10 mg/kg [Phase 2] | Dacarbazine + Intetumumab 10 mg/kg [Phase 2]
Number analyzed (Participants) | 32 | 32 | 33 | 32
Days | 54.0 [41.0 to 85.0] | 42.0 [39.0 to 43.0] | 42.0 [40.0 to 48.0] | 75.0 [43.0 to 121.0]

9. Secondary Outcome: Percentage of Participants Who Achieved a Best Overall Tumor Response as Complete Response (CR) or Partial Response (PR) - Phase 2
Description: The CR: complete disappearance of all measurable and non-measurable target lesions and PR: 50 percent (%) or more decrease in sum of the longest diameters of target lesion(s), with at least stable disease (SD) in all other evaluable disease in the absence of treatment failure. The best response achieved among all the evaluated time points was reported.
Time Frame: Screening, within 1 week of the end of Cycles 2, 4, 6, 8 (but prior to the next cycle dose), and follow-up (3 and 6 months post-last dose where applicable)
Population: The response-evaluable population included all the participants who were evaluable for response.
Measure: Number; unit: Percentage of Participants
Arm/Group | Dacarbazine + Placebo [Phase 2] | Intetumumab 5 mg/kg [Phase 2] | Intetumumab 10 mg/kg [Phase 2] | Dacarbazine + Intetumumab 10 mg/kg [Phase 2]
Number analyzed (Participants) | 31 | 31 | 33 | 30
Percentage of Participants | 9.7 | 0 | 6.1 | 3.3

10. Secondary Outcome: Percentage of Participants Who Achieved CR - Phase 2
Description: The CR: complete disappearance of all measurable and non-measurable target lesions. The participants who achieved CR as the best response were reported.
Time Frame: as for outcome 9
Population: The response-evaluable population included all the participants who were evaluable for response.
Measure: Number; unit: Percentage of Participants
Arm/Group | Dacarbazine + Placebo [Phase 2] | Intetumumab 5 mg/kg [Phase 2] | Intetumumab 10 mg/kg [Phase 2] | Dacarbazine + Intetumumab 10 mg/kg [Phase 2]
Number analyzed (Participants) | 31 | 31 | 33 | 30
Percentage of Participants | 0 | 0 | 0 | 0

11. Secondary Outcome: Percentage of Participants Who Achieved Stable Disease (SD) - Phase 2
Description: The SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for Progressive disease (PD), taking as a reference the smallest sum longest diameter since the treatment started. The participants who achieved SD as the best response were reported.
Time Frame: as for outcome 9
Population: The response-evaluable population included all the participants who were evaluable for response.
Measure: Number; unit: Percentage of Participants
Arm/Group | Dacarbazine + Placebo [Phase 2] | Intetumumab 5 mg/kg [Phase 2] | Intetumumab 10 mg/kg [Phase 2] | Dacarbazine + Intetumumab 10 mg/kg [Phase 2]
Number analyzed (Participants) | 31 | 31 | 33 | 30
Percentage of Participants | 32.3 | 25.8 | 24.2 | 53.3

12. Secondary Outcome: Overall Survival (OS) - Phase 2
Description: The OS is defined as the time from the date of randomization to the date of death due to any cause and was to be censored at the date that the subject is last known to be alive.
Time Frame: Every 3 months until death, until lost to follow-up, until withdrawal of consent, or until the Sponsor ends the study, as assessed up to 6 months post-last dose of study medication
Population: The ITT population included all the participants who were randomly assigned to treatment.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Dacarbazine + Placebo [Phase 2] | Intetumumab 5 mg/kg [Phase 2] | Intetumumab 10 mg/kg [Phase 2] | Dacarbazine + Intetumumab 10 mg/kg [Phase 2]
Number analyzed (Participants) | 32 | 32 | 33 | 32
Days | 233.0 [175.0 to 356.0] | 298.0 [213.0 to 343.0] | 426.0 [257.0 to 614.0] | 333.5 [253.0 to 536.0]

13. Secondary Outcome: Duration of Response - Phase 2
Description: Time duration required to achieve a CR or PR.
Time Frame: From the time of initial documented response (CR or PR) to the first documented sign of progression, assessed up to 6 months post-last dose of study medication
Population: The response-evaluable population included all the participants who were evaluable for response. The results were reported as individual participant's listings, but not statistically summarized.
Arm/Group | Dacarbazine + Placebo [Phase 2] | Intetumumab 5 mg/kg [Phase 2] | Intetumumab 10 mg/kg [Phase 2] | Dacarbazine + Intetumumab 10 mg/kg [Phase 2]
Number analyzed (Participants) | 0 | 0 | 0 | 0

14. Secondary Outcome: Time to Worsening in Eastern Cooperative Oncology Group (ECOG) Performance Status - Phase 2
Description: Eastern Cooperative Oncology (ECOG) performance status: Participants will be graded from 0 (Fully active, able to carry on all pre-disease activities without restriction) to 4 (Completely disabled, cannot carry on any self-care, totally confined to bed or chair). Worsening in ECOG score was defined as ≥ 1 point increase in ECOG score from baseline.
Time Frame: Baseline (within 7 days of first infusion of study medication), Day 1 of all 8 cycles, 3 weeks or 1 week post-last dose, 3 months and 6 months post-last dose of study medication
Population: The ITT population included all the participants who were randomly assigned to treatment.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Dacarbazine + Placebo [Phase 2] | Intetumumab 5 mg/kg [Phase 2] | Intetumumab 10 mg/kg [Phase 2] | Dacarbazine + Intetumumab 10 mg/kg [Phase 2]
Number analyzed (Participants) | 32 | 32 | 33 | 32
Days | 135.0 [86.0 to NA] — The upper limit of 95% confidence interval was not estimable due to inadequate events. | 226.0 [52.0 to 226.0] | 194.0 [113.0 to NA] — The upper limit of 95% confidence interval was not estimable due to inadequate events. | 170.0 [110.0 to 395.0]

15. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Intetumumab - Phase 2
Description: The maximum observed analyte concentration in serum was reported.
Time Frame: as for outcome 2
Population: The PK-evaluable population included all the participants who had at least 1 PK sample and who received at least 1 (partial or complete) dose of intetumumab.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Dacarbazine + Placebo [Phase 2] | Intetumumab 5 mg/kg [Phase 2] | Intetumumab 10 mg/kg [Phase 2] | Dacarbazine + Intetumumab 10 mg/kg [Phase 2]
Number analyzed (Participants) | 31 | 31 | 33 | 32
mcg/mL | NA (NA) — Participants in this group did not receive CNTO 95. Therefore, the data was not available for this group. | 131.18 (61.122) | 240.81 (87.332) | 219.47 (118.267)

16. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Melanoma Subscale (FACT-MS) Score - Phase 2
Description: The FACT-MS subscale is used to evaluate health related quality of life. It consists of 16 items: 12 items related to physical well-being, 3 to emotional well-being and 1 to social well-being. Scores for all items will range from 0 to 4. Total score ranges from 0-64; higher score indicates a more positive quality of life.
Time Frame: Day 1 (pre-dose) of Cycles 1, 2, 3; and final visit (3 weeks post-last dose of study medication)
Population: The ITT population included all the participants who were randomly assigned to treatment. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure and 'n' signifies those participants who were evaluable for this measure at given time points.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Dacarbazine + Placebo [Phase 2] | Intetumumab 5 mg/kg [Phase 2] | Intetumumab 10 mg/kg [Phase 2] | Dacarbazine + Intetumumab 10 mg/kg [Phase 2]
Number analyzed (Participants) | 32 | 32 | 33 | 32
Units on a scale
  Baseline (Cycle 1) (n=23, 24, 26, 26) | 53.8 (8.26) | 55.6 (5.29) | 55.3 (6.91) | 53.3 (8.22)
  Change at Cycle 2 (pre-dose) (n=20, 24, 22, 23) | -2.2 (8.13) | -1.9 (5.21) | -2.9 (5.24) | -2.0 (4.96)
  Change at Cycle 3 (pre-dose) (n = 19, 11, 5, 14) | -2.6 (7.18) | -1.3 (5.90) | 0.2 (0.84) | -0.1 (5.96)
  Change at final visit (n = 15, 20, 20, 17) | -5.7 (8.79) | -5.5 (7.08) | -2.2 (4.61) | -3.2 (8.39)

17. Secondary Outcome: Change From Baseline in Brief Pain Inventory (BPI) Score - Phase 2
Description: The BPI questionnaire is used to evaluate heath related quality of life. BPI allows participants to rate the severity of their pain on a scale of 0 (no pain) to 10 (pain as bad as you can imagine).
Time Frame: Day 1 (pre-dose) of Cycles 1, 2, 3; and final visit (3 weeks post-last dose of study medication)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Dacarbazine + Placebo [Phase 2] | Intetumumab 5 mg/kg [Phase 2] | Intetumumab 10 mg/kg [Phase 2] | Dacarbazine + Intetumumab 10 mg/kg [Phase 2]
Number analyzed (Participants) | 32 | 32 | 33 | 32
Units on a scale
  Baseline (Cycle 1) (n=23, 23, 27, 25) | 1.3 (1.77) | 2.0 (2.50) | 0.9 (1.79) | 2.2 (2.37)
  Change at Cycle 2 (pre-dose) (n=20, 22, 22, 22) | 0.9 (1.92) | 0.0 (1.96) | 0.5 (2.09) | -0.3 (1.94)
  Change at Cycle 3 (pre-dose) (n = 19, 10, 6, 14) | 0.5 (2.41) | 0.5 (1.27) | 0.0 (0.63) | -0.8 (2.19)
  Change at final visit (n = 15, 20, 20, 16) | 1.4 (2.85) | 0.8 (1.80) | 1.0 (1.96) | 0.3 (3.48)

18. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Intetumumab - Phase 1 (Part 2)
Description: The maximum observed analyte concentration in serum was reported.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Microgram per milliliter (mcg/mL)
Arm/Group | Dacarbazine + Intetumumab 5 mg/kg [Phase 1 (Part 2)] | Dacarbazine + Intetumumab 10 mg/kg [Phase 1 (Part 2)]
Number analyzed (Participants) | 3 | 2
Microgram per milliliter (mcg/mL) | 118.47 (33.462) | 220.87 (122.662)

19. Secondary Outcome: Area Under the Serum Concentration Versus Time Curve (AUC) of Intetumumab - Phase 1 (Part 2)
Description: The AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mcg*day/mL
Arm/Group | Dacarbazine + Intetumumab 5 mg/kg [Phase 1 (Part 2)] | Dacarbazine + Intetumumab 10 mg/kg [Phase 1 (Part 2)]
Number analyzed (Participants) | 2 | 1
mcg*day/mL | 368.74 (36.056) | 963.17 (NA) — Standard deviation was not estimable based on one subject.

20. Secondary Outcome: Half-life of Intetumumab - Phase 1 (Part 2)
Description: Plasma decay half-life is the time measured for the plasma concentration of the drug to decrease by one half.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Dacarbazine + Intetumumab 5 mg/kg [Phase 1 (Part 2)] | Dacarbazine + Intetumumab 10 mg/kg [Phase 1 (Part 2)]
Number analyzed (Participants) | 2 | 1
Days | 2.41 (0.559) | 2.36 (NA) — Standard deviation was not estimable based on one subject.

21. Secondary Outcome: Total Clearance (CL) of Intetumumab After Intravenous Administration - Phase 1 (Part 2)
Description: The CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/day/kg
Arm/Group | Dacarbazine + Intetumumab 5 mg/kg [Phase 1 (Part 2)] | Dacarbazine + Intetumumab 10 mg/kg [Phase 1 (Part 2)]
Number analyzed (Participants) | 2 | 1
mL/day/kg | 13.44 (1.537) | 10.34 (NA) — Standard deviation was not estimable based on one subject.

22. Secondary Outcome: Volume of Distribution (Vz) of Intetumumab - Phase 1 (Part 2)
Description: as for outcome 6
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | Dacarbazine + Intetumumab 5 mg/kg [Phase 1 (Part 2)] | Dacarbazine + Intetumumab 10 mg/kg [Phase 1 (Part 2)]
Number analyzed (Participants) | 2 | 1
mL/kg | 47.38 (16.187) | 35.18 (NA) — Standard deviation was not estimable based on one subject.

23. Secondary Outcome: Accumulation Ratio (R) of Intetumumab - Phase 1 (Part 2)
Description: The R is obtained by dividing AUC at two different time points.
Time Frame: as for outcome 2
Population: as for outcome 7
Arm/Group | Dacarbazine + Intetumumab 5 mg/kg [Phase 1 (Part 2)] | Dacarbazine + Intetumumab 10 mg/kg [Phase 1 (Part 2)]
Number analyzed (Participants) | 0 | 0

24. Other Pre Specified Outcome: Area Under the Concentration Versus Time Curve Between Zero to Infinite Time (AUCinf) of Intetumumab - Phase 1 (Part 1)
Description: The AUCinf = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mcg*day/mL
Arm/Group | Intetumumab 3 mg/kg [Phase 1 (Part 1)] | Intetumumab 5 mg/kg [Phase 1 (Part 1)] | Intetumumab 10 mg/kg [Phase 1 (Part 1)]
Number analyzed (Participants) | 1 | 1 | 3
mcg*day/mL | 257.80 (NA) — Standard deviation was not estimable based on one subject. | 503.88 (NA) — Standard deviation was not estimable based on one subject. | 1591.54 (213.858)

25. Other Pre Specified Outcome: Percentage of Participants Who Achieved a Best Overall Response as CR, PR, or SD - Phase 2
Description: The CR: complete disappearance of all measurable and non-measurable target lesions and PR: 50% or more decrease in sum of the longest diameters of target lesion(s), with at least stable disease (SD) in all other evaluable disease in the absence of treatment failure.
Time Frame: Within 28 days of first infusion of study medication, within 1 week of the end of Cycles 2, 4, 6, 8; 3 months and 6 months post-last dose of study medication
Population: The response-evaluable population included all the participants who were evaluable for response.
Measure: Number; unit: Percentage of Participants
Arm/Group | Dacarbazine + Placebo [Phase 2] | Intetumumab 5 mg/kg [Phase 2] | Intetumumab 10 mg/kg [Phase 2] | Dacarbazine + Intetumumab 10 mg/kg [Phase 2]
Number analyzed (Participants) | 31 | 31 | 33 | 30
Percentage of Participants | 41.9 | 25.8 | 30.3 | 56.7

ADVERSE EVENTS:
Time Frame: Day 1 up to Follow-up period (30 days post-last dose).
Arm/Group | Intetumumab 3 mg/kg [Phase 1 (Part 1)] | Intetumumab 5 mg/kg [Phase 1 (Part 1)] | Intetumumab 10 mg/kg [Phase 1 (Part 1)] | Dacarbazine + Intetumumab 5 mg/kg [Phase 1 (Part 2)] | Dacarbazine + Intetumumab 10 mg/kg [Phase 1 (Part 2)] | Dacarbazine + Placebo [Phase 2] | Intetumumab 5 mg/kg [Phase 2] | Intetumumab 10 mg/kg [Phase 2] | Dacarbazine + Intetumumab 10 mg/kg [Phase 2]
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 0/3 | 1/3 | 2/3 | 9/31 | 4/31 | 6/33 | 7/32
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 2/3 | 3/3 | 3/3 | 30/31 | 30/31 | 32/33 | 30/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intetumumab 3 mg/kg [Phase 1 (Part 1)] (N=3) | Intetumumab 5 mg/kg [Phase 1 (Part 1)] (N=3) | Intetumumab 10 mg/kg [Phase 1 (Part 1)] (N=3) | Dacarbazine + Intetumumab 5 mg/kg [Phase 1 (Part 2)] (N=3) | Dacarbazine + Intetumumab 10 mg/kg [Phase 1 (Part 2)] (N=3) | Dacarbazine + Placebo [Phase 2] (N=31) | Intetumumab 5 mg/kg [Phase 2] (N=31) | Intetumumab 10 mg/kg [Phase 2] (N=33) | Dacarbazine + Intetumumab 10 mg/kg [Phase 2] (N=32)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Cyanosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye Haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Disease Progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
General Physical Health Deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Anaphylactic Reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis Norovirus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malignant Pleural Effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Metastases to Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin Neoplasm Bleeding (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypotonia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Reversible Posterior Leukoencephalopathy Syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal Cord Compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pallor (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intetumumab 3 mg/kg [Phase 1 (Part 1)] (N=3) | Intetumumab 5 mg/kg [Phase 1 (Part 1)] (N=3) | Intetumumab 10 mg/kg [Phase 1 (Part 1)] (N=3) | Dacarbazine + Intetumumab 5 mg/kg [Phase 1 (Part 2)] (N=3) | Dacarbazine + Intetumumab 10 mg/kg [Phase 1 (Part 2)] (N=3) | Dacarbazine + Placebo [Phase 2] (N=31) | Intetumumab 5 mg/kg [Phase 2] (N=31) | Intetumumab 10 mg/kg [Phase 2] (N=33) | Dacarbazine + Intetumumab 10 mg/kg [Phase 2] (N=32)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 1 | 0 | 6 | 1 | 0 | 7
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 6
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 0 | 7 | 0 | 0 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 8 | 0 | 0 | 6
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye Irritation (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye Pain (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0
Lacrimation Increased (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ocular Discomfort (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ocular Hyperaemia (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uveitis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 7 | 10 | 7
Visual Acuity Reduced (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous Floaters (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 2
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 1
Abdominal Tenderness (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 2 | 6 | 3 | 3 | 7
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 3 | 3 | 6 | 7
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 0 | 1 | 0 | 16 | 7 | 12 | 15
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 4 | 6 | 13 | 8
Chest Pain (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Chills (General disorders) | 1 | 3 | 0 | 1 | 1 | 5 | 5 | 9 | 5
Fatigue (General disorders) | 2 | 2 | 0 | 3 | 1 | 13 | 7 | 14 | 10
Influenza Like Illness (General disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 5 | 3 | 2
Infusion Site Extravasation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion Site Pain (General disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 6
Oedema Peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 3 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 5 | 1 | 1
Pyrexia (General disorders) | 2 | 3 | 0 | 0 | 1 | 4 | 9 | 12 | 6
Abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1
Oral Herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Wound Secretion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Blood Creatinine Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Blood Lactate Dehydrogenase Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0
Heart Rate Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Weight Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 4 | 0 | 4
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1 | 0 | 2 | 1 | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 3 | 1
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 5
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1
Disturbance in Attention (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 2
Headache (Nervous system disorders) | 3 | 3 | 2 | 2 | 2 | 12 | 16 | 23 | 12
Neuropathy Peripheral (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 3
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Libido Decreased (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Menstruation Irregular (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sexual Dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1 | 0 | 3 | 0 | 5 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 1 | 6 | 3 | 1 | 5
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hot Flush (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less